CLINICAL TRIAL: NCT04698187
Title: A Multicenter, Open-label, Phase 2 Study of Intratumoral CMP-001 in Combination With Intravenous Nivolumab in Subjects With Refractory Unresectable or Metastatic Melanoma
Brief Title: CMP-001 in Combination With Nivolumab in Subjects With Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMP-001-010
Record Dates: First submitted 2020-12-10; First posted 2021-01-06 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Melanoma; Advanced Melanoma; Metastatic Melanoma; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CMP-001 and Nivolumab (Experimental): All enrolled subjects will receive CMP-001 IT and nivolumab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: CMP-001; Drug: Nivolumab

INTERVENTIONS:
Drug: CMP-001 — Subjects will receive CMP-001 10 mg IT weekly for 7 doses after which CMP-001 will be administered every 3 weeks (Q3W).
  Other Names: vidutolimod
Drug: Nivolumab — Nivolumab 360 mg IV is administered Q3W.
  Other Names: OPDIVO

SUMMARY:
CMP-001-010 is a Phase 2 study of CMP-001 intratumoral (IT) and nivolumab intravenous (IV) administered to participants with refractory unresectable or metastatic melanoma.

The primary objective of the study is to determine confirmed objective response with CMP-001 in combination with nivolumab in subjects with refractory unresectable or metastatic melanoma.

The secondary objectives are to:

* To evaluate the safety and tolerability of CMP-001 administered by intratumoral (IT) injection in combination with nivolumab in subjects with refractory unresectable or metastatic melanoma.
* To evaluate the efficacy of CMP-001 in combination with nivolumab in subjects with refractory unresectable or metastatic melanoma.
* To assess the pharmacokinetic (PK) profile of CMP-001 in combination with nivolumab in subjects with refractory unresectable or metastatic melanoma.
* To assess and describe the immunogenicity of CMP-001 in combination with nivolumab in subjects with refractory unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
Former Sponsor Checkmate Pharmaceuticals

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the study must meet all of the following inclusion criteria to be eligible.

1. Histopathologically-confirmed diagnosis of malignant melanoma that is metastatic or unresectable at Screening.
2. Known BRAF mutation status; if BRAF V600 mutation positive, must have had prior treatment with a local Health Authority approved BRAF inhibitor, with or without mitogen-activated protein kinase inhibitor. Patients with BRAF V600 mutations who refuse a BRAF inhibitor will not be eligible.
3. Refractory to PD-1 blockade either as monotherapy or in combination with other therapies, as defined by the following criteria:

   1. Received treatment with a Food and Drug Administration approved PD-1 blocking antibody for 12 weeks or longer.
   2. Have PD (according to RECIST v1.1) within 12 weeks of the last dose of a PD-1 blocking antibody, either as monotherapy or in combination with other agents.

   Evidence of confirmed PD must be established by investigator assessment at least 4 weeks after the initial date of PD. The second assessment may serve as the Baseline for this study if completed within 30 days before to the start of study treatment. NOTE: in subjects with histologically confirmed recurrence on or after adjuvant PD-1 blocking antibody, confirmatory imaging is not required.
4. Measurable disease, as defined by RECIST v1.1 and all of the following:

   1. At least 1 accessible lesion amenable to repeated IT injection.
   2. One or more measurable lesions at least 1 cm in diameter that are not intended for CMP 001 injection and can be followed as target lesions per RECIST v1.1.
   3. Documented disease progression in any lesion that was previously radiated in order to serve as a target lesion.
5. Able to provide tissue from a core or excisional biopsy (fine needle aspirate is not sufficient). A fresh tissue biopsy (within 90 days before the start of study treatment) is preferred but an archival sample is acceptable if no intervening therapy was received. Note: For tissue sampling details, please refer to the laboratory manual.
6. Adequate organ function based on most recent laboratory values within 3 weeks before first dose of study treatment on Week 1 Day 1 (W1D1):

   1. Bone marrow function:

      * neutrophil count ≥ 1500/mm3
      * platelet count ≥ 100,000/mm3
      * hemoglobin concentration ≥ 9 g/dL
      * white blood cells ≥ 2000/mm3
   2. Liver function:

      * total bilirubin ≤ 1.5 times the upper limit of normal (ULN) with the following exception: patients with Gilbert Disease total serum bilirubin ≤ 3 times ULN
      * aspartate aminotransferase and alanine aminotransferase ≤ 3 times the ULN
   3. Lactate dehydrogenase ≤ 2 times the ULN
   4. Renal function: estimated (Cockcroft-Gault) or measured creatinine clearance ≥ 30 mL/min.
   5. Coagulation:

      * International normalized ratio or prothrombin time (PT) ≤ 1.5 times ULN, unless subject is receiving anticoagulant therapy, as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
      * Activated partial thromboplastin time or PTT ≤ 1.5 times ULN, unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
7. Age ≥ 18 years at time of consent.
8. Eastern Cooperative Oncology Group Performance Status of 0 to 1 at Screening.
9. Capable of understanding and complying with protocol requirements.
10. Women of childbearing potential must have negative serum pregnancy test before dosing at W1D1 and be willing to use an adequate method of contraception from the time of consent until at least 150 days after last dose of study treatment.
11. Able and willing to provide written informed consent and to follow study instructions. Subjects unable to provide written informed consent on their own behalf will not be eligible for the study.

Exclusion Criteria:

Subjects presenting with any of the following will not qualify for entry into the study:

1. Uveal, acral, or mucosal melanoma.
2. Received radiation therapy (or other nonsystemic therapy) within 2 weeks before first dose of study treatment on W1D1. Patients should have recovered (ie, Grade ≤1 or at baseline) from radiation-related toxicities.
3. Treatment with complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before start of study treatment. Refer to Section 4.4. for prohibited therapies.
4. Received systemic pharmacologic doses of corticosteroids ≥10 mg/day prednisone within 30 days before first dose of study treatment on W1D1.

   1. Subjects who are currently receiving steroids at a prednisone-equivalent dose of ≤ 10 mg/day do not need to discontinue steroids before enrollment.
   2. Replacement doses, topical, ophthalmologic, and inhalational steroids are permitted.
   3. Stress-dose corticosteroids will be required in subjects with adrenal insufficiency
5. History of immune-related AE that required permanent discontinuation of PD-1 blocking antibody.
6. Not fully recovered from AEs (to Grade 1 or less [per CTCAE v5.0], with the exception of persistent adverse events or sequelae, eg, vitiligo, alopecia, hypothyroidism, diabetes mellitus, and adrenal and/or pituitary insufficiency) due to prior treatment.

   NOTE: Subjects previously treated with a CTLA-4-blocking antibody, subjects receiving corticosteroids with daily doses > 5 mg and ≤ 10 mg of prednisone equivalent for 2 weeks, and subjects with clinical symptoms and/or laboratory findings suggesting risk for adrenal insufficiency should undergo diagnostic tests for adrenal insufficiency via local laboratory.
7. Active pneumonitis or history of noninfectious pneumonitis that required steroids.
8. Severe uncontrolled cardiac disease within 6 months of Screening, including but not limited to poorly controlled hypertension, unstable angina, myocardial infarction, congestive heart failure (New York Heart Association Class II or greater), pericarditis within the previous 6 months, cerebrovascular accident, or implanted or continuous use of a pacemaker or defibrillator.
9. Known history of immunodeficiency.
10. Known additional malignancy that is progressing or required active treatment within the past 3 years. Exceptions include cancers that have undergone potentially curative therapy, eg, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, localized prostate cancer with prostate-specific antigen level below 4.0 ng/mL, in situ cervical cancer on biopsy or a squamous intraepithelial lesion on Papanicolaou smear, and thyroid cancer (except anaplastic), in situ breast cancer, and adjuvant hormonal therapy for breast cancer > 3 years from curative-intent surgical resection.
11. Active autoimmune disease that has required systemic treatment in past 2 years; replacement therapy is not considered a form of systemic treatment.
12. Untreated, symptomatic, or enlarging central nervous system metastases or carcinomatous meningitis (including leptomeningeal metastases from solid tumors).
13. Prior allogenic tissue/solid organ transplant.
14. Active infection requiring systemic therapy.
15. Known or suspected active infection with severe acute respiratory syndrome coronavirus 2 virus.
16. Known or suspected active infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus (testing is not required unless suspected).
17. Received a live virus/attenuated vaccination within 30 days before first dose of study treatment on W1D1.
18. Received blood products (including platelets or red blood cells) or colony stimulating factors (including granulocyte colony stimulating factor, granulocyte/macrophage colony stimulating factor, or recombinant erythropoietin) within 30 days before the start of Screening.
19. History of allergy or hypersensitivity to nivolumab and/or any of its excipients.
20. Any concurrent uncontrolled illness, including mental illness or substance abuse, which in the opinion of the Investigator would make the subject unable to cooperate or participate in the study.
21. Participation in another clinical study of an investigational anticancer therapy or device within 30 days before first dose of study treatment on W1D1. Participation in the follow-up phase (receiving no study treatment) of a prior study is allowed.
22. Requires prohibited treatment (ie, non-protocol specified anticancer pharmacotherapy, surgery, or radiotherapy) for treatment of malignant tumor.
23. Has a life expectancy of less than 3 months and/or has rapidly progressing disease (eg, tumor bleeding, uncontrolled tumor pain) in the opinion of the treating Investigator.
24. Received previous CMP-001 treatment.
25. Pregnant or breastfeeding or expecting to conceive or donate eggs within the projected duration of the study, from the time of consent until at least 150 days after last dose of study treatment for women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (25):
- United States (25):
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope National Medical Center, Robert Kang, MD, Duarte, California
  - UCLA Hematology-Oncology, Los Angeles, California
  - California Cancer Associates for Research & Excellence, Inc., San Marcos, California
  - University of Colorado- Denver, Denver, Colorado
  - Hartford Healthcare, Hartford, Connecticut
  - GenesisCare USA, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Louisville Health Care, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Cancer Institute, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sammons Cancer Center, Dallas, Texas
  - University of Utah- Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- CMP-001 + Nivolumab: All participants received CMP-001 intratumorally (IT) and nivolumab intravenously (IV) according to the treatment schedule.
Period: Overall Study
Arm/Group | CMP-001 + Nivolumab
Started (Received at least 1 dose of study treatment) | 44
Completed | 0
Not Completed | 44
Not completed — Withdrawal by Subject | 7
Not completed — Death | 21
Not completed — Sponsor Decision | 15
Not completed — In-transit Disease | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set (includes all participants who received at least 1 [partial or full] dose of study treatment)
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (14.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 41
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) by Blinded Independent Central Review (BICR)
Description: ORR, defined as the percentage of participants who have confirmed best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as assessed by Blinded Independent Central Review (BICR)
Time Frame: Up to approximately 24 months (107 weeks)
Population: Intent-to-Treat (ITT) Analysis Set (included all participants who received at least 1 [partial or full] dose of study treatment)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 44
Percentage of participants | 11.4 [3.79 to 24.56]

2. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Any Serious TEAE, and Any TEAE Leading to Discontinuation or Death
Description: Number of participants with any treatment-emergent adverse event (TEAE), any serious TEAE, and any TEAE leading to discontinuation or death reported.
Time Frame: Up to approximately 24 months (107 weeks)
Population: Safety Analysis Set (all participants who received at least 1 dose of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 44
Participants
  Any TEAE | 44
  Any serious TEAE | 12
  Any TEAE leading to death | 1

3. Secondary Outcome: Severity of TEAEs as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Description: Number of participants per NCI CTCAE version 5.0 Adverse Event Grade reported:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2 Moderate; minimal, local, or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limited self-care activities of daily living Grade 4 Life-threatening consequences: urgent intervention indicated Grade 5 Death related to adverse event
Time Frame: Up to approximately 24 months (107 weeks)
Population: Safety Analysis Set (all participants who received at least 1 dose of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 44
Participants
  Grade 1 Mild | 2
  Grade 2 Moderate | 18
  Grade 3 Severe | 21
  Grade 4 Life-threatening | 2
  Grade 5 Death | 1

4. Secondary Outcome: Time to Response (TTR) by BICR
Description: TTR, defined as the time from the first dose date of the study treatment to the first time when criteria are first met for CR or PR, whichever occurred first, per RECIST v1.1 by BICR.
Time Frame: Up to approximately 28 months (122 weeks)
Population: Number of participants analyzed for TTR included only participants who had a confirmed best overall response (BOR) of complete response (CR) or partial response (PR).
Measure: Median (Full Range); unit: Months
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 5
Months | 2.89 [2.69 to 5.32]

5. Secondary Outcome: Time to Response (TTR) by Investigator
Description: TTR, defined as the time from the first dose date of the study treatment to the first time when criteria are first met for CR or PR, whichever occurred first, per RECIST v1.1 by Investigator.
Time Frame: Up to approximately 28 months (122 weeks)
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 7
Months | 2.89 [2.53 to 4.86]

6. Secondary Outcome: Duration of Response (DOR) by BICR
Description: DOR, defined as time from the date of first documented response (CR or PR) to the date of documented progressive disease (PD), based on RECIST v1.1 by BICR.
Time Frame: Up to approximately 28 months (122 weeks)
Population: Number of participants analyzed for DOR included only participants who had a confirmed best overall response (BOR) of complete response (CR) or partial response (PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 5
Months | NA [3.351 to NA] — Insufficient number of participants with events

7. Secondary Outcome: Duration of Response (DOR) by Investigator
Description: DOR, defined as time from the date of first documented response (CR or PR) to the date of documented progressive disease (PD), based on RECIST v1.1 by Investigator.
Time Frame: Up to approximately 28 months (122 weeks)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 7
Months | NA [3.351 to NA] — Insufficient number of participants with events

8. Secondary Outcome: Confirmed ORR in Non-injected Target Lesions by Investigator
Description: Confirmed ORR, defined as the percentage of participants in the analysis set who had confirmed BOR of CR or PR based on RECIST v1.1 as assessed by Investigator.
Time Frame: Up to approximately 24 months (107 weeks)
Population: Number of participants analyzed included only participants who had at least one non-injected target lesion.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 43
Percentage of participants | 16.3 [6.81 to 30.70]

9. Secondary Outcome: Progression-free Survival (PFS) by BICR
Description: PFS, defined as time from date of first dose of study treatment to date of documented PD based on RECIST v1.1 by BICR or death, whichever occurred first.
Time Frame: Up to approximately 31 months (135 weeks)
Population: ITT Analysis Set (included all participants who received at least 1 [partial or full] dose of study treatment)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 44
Months | 2.83 [2.595 to 4.731]

10. Secondary Outcome: Progression-free Survival (PFS) by Investigator
Description: PFS, defined as time from date of first dose of study treatment to date of documented PD based on RECIST v1.1 by Investigator or death, whichever occurred first.
Time Frame: Up to approximately 31 months (135 weeks)
Population: ITT Analysis Set (included all participants who received at least 1 [partial or full] dose of study treatment)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 44
Months | 2.79 [2.628 to 4.172]

11. Secondary Outcome: Overall Survival (OS) by Investigator
Description: OS, defined as the time from the first dose date of the study treatment to the date of death from any cause.
Time Frame: Up to approximately 32 months (139 weeks)
Population: ITT Analysis Set (included all participants who received at least 1 [partial or full] dose of study treatment)
Measure: Median (Full Range); unit: Months
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 44
Months | 18.43 [0.76 to 31.93]

12. Secondary Outcome: Immune Objective Response Rate (iORR) by Investigator
Description: iORR, defined as the percentage of participants with an immune best overall response (iBOR) of confirmed immune complete response (iCR) or confirmed immune partial response (iPR) based on immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) by Investigator assessment.
Time Frame: Up to approximately 24 months (107 weeks)
Population: iORR is only defined for participants who continued study treatment beyond progressive disease (PD) per RECIST v1.1 as assessed by the Investigator according to immunotherapy RECIST (iRECIST). Here, 6 participants met the criteria for iORR assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 6
Percentage of Participants | NA — Insufficient number of participants with immune response

13. Secondary Outcome: Immune Duration of Response (iDOR) by Investigator
Description: iDOR, defined as the time from the date of the first immune response (iCR or iPR) to the date of immune confirmed progressive disease (iCPD) by Investigator assessment.
Time Frame: Up to approximately 28 months (122 weeks)
Population: iDOR is only defined for participants who had a confirmed iBOR of iCR or iPR. Here, 0 participants met the criteria.
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Immune Progression-free Survival (iPFS) by Investigator
Description: iPFS, defined as the time from the first dose date of the study treatment to date of immune confirmed progressive disease (iCPD) per iRECIST by Investigator assessment or death, whichever occurred first.
Time Frame: Up to 9 months (approximately 39 weeks)
Population: ITT Analysis Set (included all participants who received at least 1 [partial or full] dose of study treatment)
Measure: Median (Full Range); unit: Months
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 44
Months | 8.542 [0.03 to 9.00]

15. Secondary Outcome: Maximum Observed Serum Concentration
Description: Assess the pharmacokinetic (PK) profile for maximum observed serum concentration.
Time Frame: From first dose of drug (Week 1 Day 1) until 30 days after the last drug injection (until a reason for treatment discontinuation occurs)
Population: Per protocol, the pharmacokinetic (PK) Analysis Set was defined as all participants who received CMP-001 and had evaluable serum samples at Baseline and after CMP-001 injection. Here, no participants had evaluable serum samples at any time therefore, Number of Participants Analyzed equals 0.
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 0

16. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to the Last Quantifiable Time Point
Description: Assess the PK profile for area under the serum concentration-time curve from time zero to the last quantifiable time point.
Time Frame: as for outcome 15
Population: as for outcome 15
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 0

17. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity
Description: Assess the PK profile for area under the serum concentration-time curve from time zero extrapolated to infinity.
Time Frame: as for outcome 15
Population: as for outcome 15
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 0

18. Secondary Outcome: Terminal Elimination Half-Life
Description: Assess the PK profile for terminal elimination half-life.
Time Frame: as for outcome 15
Population: as for outcome 15
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 0

19. Secondary Outcome: Number of Participants With Immunogenicity as Measured by Anti-Qbeta Antibodies (ADA)
Description: Development of anti-Qbeta antibodies in participants with refractory unresectable or metastatic melanoma.
Time Frame: Up to approximately 24 months (107 weeks)
Population: The Immunogenicity Analysis Set is defined as all participants who received at least 1 dose of CMP-001 and have at least 1 non-missing ADA result after CMP-001 administration.
Measure: Count of Participants; unit: Participants
Arm/Group | CMP-001 + Nivolumab
Number analyzed (Participants) | 41
Participants | 41

ADVERSE EVENTS:
Time Frame: From signing of informed consent through end of study up to approximately 32 months (139 weeks).
Arm/Group | CMP-001 + Nivolumab
All-Cause Mortality (participants affected / at risk) | 21/44
Serious Adverse Events (participants affected / at risk) | 12/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMP-001 + Nivolumab (N=44)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMP-001 + Nivolumab (N=44)
Fatigue (General disorders) | 21 (40)
Chills (General disorders) | 20 (51)
Pyrexia (General disorders) | 20 (43)
Injection site erythema (General disorders) | 9 (9)
Injection site pain (General disorders) | 9 (10)
Oedema peripheral (General disorders) | 7 (11)
Influenza like illness (General disorders) | 5 (16)
Chest discomfort (General disorders) | 3 (4)
Injection site reaction (General disorders) | 3 (3)
Injection site swelling (General disorders) | 3 (3)
Localised oedema (General disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 17 (25)
Vomiting (Gastrointestinal disorders) | 16 (23)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Hypotension (Vascular disorders) | 15 (31)
Hypertension (Vascular disorders) | 7 (21)
Flushing (Vascular disorders) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (14)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4)
Lipase increased (Investigations) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 5 (7)
Blood lactate dehydrogenase increased (Investigations) | 4 (10)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3)
Amylase increased (Investigations) | 3 (4)
Blood creatinine increased (Investigations) | 3 (4)
Lymphocyte count decreased (Investigations) | 3 (4)
Neutrophil count decreased (Investigations) | 3 (13)
Weight decreased (Investigations) | 3 (4)
Weight increased (Investigations) | 3 (3)
Headache (Nervous system disorders) | 12 (19)
Dizziness (Nervous system disorders) | 8 (9)
Anaemia (Blood and lymphatic system disorders) | 13 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8)
COVID-19 (Infections and infestations) | 5 (6)
Skin infection (Infections and infestations) | 3 (4)
Tachycardia (Cardiac disorders) | 4 (7)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (8)

LIMITATIONS AND CAVEATS:
The study stopped before reaching sample size as originally planned (n=100) for analysis per protocol. This was a business decision independent of safety/efficacy findings. Assessment of PK was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT04698187/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT04698187/SAP_001.pdf